CLINICAL TRIAL: NCT03930953
Title: A Phase 1/2, Multi-center, Open-label Study to Assess the Safety, Pharmacokinetics, and Preliminary Efficacy of an Orally Available Small Molecule, CC-99282, Alone and in Combination With Anti-Lymphoma Agents in Subjects With Relapsed or Refractory Non-Hodgkin Lymphomas (R/R NHL).
Brief Title: A Safety and Preliminary Efficacy Study of CC-99282, Alone and in Combination With Anti-lymphoma Agents in Participants With Relapsed or Refractory Non-Hodgkin Lymphomas (R/R NHL)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CC-99282-NHL-001; U1111-1224-5399 (Registry Identifier: WHO); 2018-003235-29 (EudraCT Number)
Record Dates: First submitted 2019-04-16; First posted 2019-04-29 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Non-Hodgkin Lymphomas (NHL); Safety; Efficacy; CC-99282; Rituximab; Relapsed; Refractory; Pharmacokinetics; Obinutuzumab; Tafasitamab; Valemetostat; Anti-lymphoma agents
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence | interventions — Rituximab; obinutuzumab; tafasitamab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: Dose Escalation (Experimental)
  Interventions: Drug: CC-99282
- Part B: Dose Expansion (Experimental)
  Interventions: Drug: CC-99282; Drug: Rituximab; Drug: Obinutuzumab; Drug: Tafasitamab; Drug: Valemetostat

INTERVENTIONS:
Drug: CC-99282 — Specified dose on specified days
  Other Names: BMS-986369
Drug: Rituximab — Specified dose on specified days
  Arms: Part B: Dose Expansion
Drug: Obinutuzumab — Specified dose on specified days
  Arms: Part B: Dose Expansion
Drug: Tafasitamab — Specified dose on specified days
  Arms: Part B: Dose Expansion
Drug: Valemetostat — Specified dose on specified days
  Arms: Part B: Dose Expansion

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and preliminary efficacy of CC-99282 alone and in combination with anti-lymphoma agents in participants with relapsed or refractory non-Hodgkin's lymphomas.

DETAILED DESCRIPTION:
Participants with relapsed or refractory non-Hodgkin's lymphomas (R/R NHL) who have failed at least 2 lines of therapy (or have received at least one prior line of standard therapy and are not eligible for any other therapy).

The dose escalation will evaluate the safety and tolerability of escalating doses of CC-99282 in relapsed or refractory diffuse large B-cell lymphoma (R/R DLBCL) and/or relapsed or refractory follicular lymphoma (R/R FL) participants to determine the maximum tolerated dose (MTD) of CC-99282 as monotherapy.

The dose expansion will further evaluate the safety and preliminary efficacy of single agent CC-99282 or the safety and preliminary efficacy of CC-99282 in combination with anti-lymphoma agents in participants with R/R DLBCL and NHL.

Part B Cohort B will further evaluate the potential effects of food on the PK and safety of CC-99282.

ELIGIBILITY:
Inclusion Criteria:

* History of Non-Hodgkin's Lymphoma (NHL) with relapsed or refractory disease
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2

Exclusion Criteria:

* Life expectancy ≤ 2 months
* Received prior systemic anti-cancer treatment (approved or investigational) ≤ 5 half-lives or 4 weeks prior to starting CC-99282, whichever is shorter
* Is on chronic systemic immunosuppressive therapy or corticosteroids or has clinically significant graft-versus-host disease (GVHD)
* Impaired cardiac function or clinically significant cardiac disease

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2027-04-07 (Estimated); Study Completion 2028-02-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) | From the time of consent at screening until 28 days after the subject discontinued study treatment (up to 4 years)
Number of participants with laboratory abnormalities | From the time of consent at screening until 28 days after the subject discontinued study treatment (up to 4 years)
Number of participants with vital sign abnormalities | From the time of consent at screening until 28 days after the subject discontinued study treatment (up to 4 years)
Number of participants with electrocardiogram (ECG) abnormalities | From the time of consent at screening until 28 days after the subject discontinued study treatment (up to 4 years)
Number of participants with Eastern Cooperative Oncology Group (ECOG) performance status abnormalities | From the time of consent at screening until 28 days after the subject discontinued study treatment (up to 4 years)
Number of participants with left ventricular ejection fraction (LVEF) assessment abnormalities | From the time of consent at screening until 28 days after the subject discontinued study treatment (up to 4 years)
Number of participants with physical examination abnormalities | From the time of consent at screening until 28 days after the subject discontinued study treatment (up to 4 years)
Dose Limiting Toxicity (DLT) | Up to 28 days in Cycle 1
Maximum tolerated dose (MTD) | Up to 28 days in cycle 1

SECONDARY OUTCOMES:
Pharmacokinetics - Maximum plasma concentration of drug (Cmax) | Cycle 1 to Cycle 4 Day 15 (each cycle is 28 days)
Pharmacokinetics - Area under the plasma concentration-time curve (AUC) | Cycle 1 to Cycle 4 Day 15 (each cycle is 28 days)
Pharmacokinetics - Time to peak (maximum) plasma concentration (Tmax) | Cycle 1 to Cycle 4 Day 15 (each cycle is 28 days)
Pharmacokinetics - Terminal-phase elimination half-life (T-HALF) | Cycle 1 to Cycle 4 Day 15 (each cycle is 28 days)
Pharmacokinetics - Apparent total body clearance of the drug from the plasma (CLT/F) | Cycle 1 to Cycle 4 Day 15 (each cycle is 28 days)
Pharmacokinetics: Apparent volume of distribution (Vz/F) | Cycle 1 to Cycle 4 Day 15 (each cycle is 28 days)
Objective response rate (ORR) | Up to approximately 6 years
  Defined as the percent of subjects whose best response is Complete Response (CR) or Partial Response (PR).
  Determined by the Lugano Classification for NHL response criteria
Time to response (TTR) | Up to approximately 6 years
  Determined by the Lugano Classification for NHL response criteria
Duration of response (DoR) | Up to approximately 6 years
  Determined by the Lugano Classification for NHL response criteria
Progression free survival (PFS) | Up to approximately 6 years
  Time from first dose of CC-99282 to the first occurrence of disease progression or death from any cause
  Determined by the Lugano Classification for NHL response criteria
Overall survival (OS) | Up to approximately 6 years
  Time from first dose of CC-99282 to death from any cause
  Determined by the Lugano Classification for NHL response criteria
ORR | Up to approximately 4 years
  Defined as the percent of subjects whose best response is Complete Response (CR) or Partial Response (PR).
  Determined using the modified International PCNSL Collaborative Group (IPCG) criteria
TTR | Up to approximately 4 years
  Determined using the modified International PCNSL Collaborative Group (IPCG) criteria
DOR | Up to approximately 4 years
  Determined using the modified International PCNSL Collaborative Group (IPCG) criteria
PFS | Up to approximately 4 years
  Determined using the modified International PCNSL Collaborative Group (IPCG) criteria
OS | Up to approximately 4 years
  Determined using the modified International PCNSL Collaborative Group (IPCG) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (66):
- United States (8):
  - Local Institution - 109, Scottsdale, Arizona
  - Local Institution - 111, Jacksonville, Florida
  - Local Institution - 102, Tampa, Florida
  - Local Institution - 108, Overland Park, Kansas
  - Local Institution - 107, Rochester, Minnesota
  - Local Institution - 104, St Louis, Missouri
  - Local Institution - 103, Hackensack, New Jersey
  - Local Institution - 101, Houston, Texas
- Argentina (3):
  - Local Institution - 255, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Local Institution - 254, Pilar, Buenos Aires
  - Local Institution - 253, Buenos Aires
- Austria (3):
  - Local Institution - 701, Salzburg
  - Local Institution - 704, Sankt Pölten
  - Local Institution - 703, Vienna
- Local Institution - 902, Leuven, Belgium
- Brazil (4):
  - Local Institution - 453, Porto Alegre, Rio Grande do Sul
  - Local Institution - 450, São Paulo, São Paulo
  - Local Institution - 451, São Paulo
  - Local Institution - 452, São Paulo
- Local Institution - 201, Toronto, Ontario, Canada
- Chile (5):
  - Local Institution - 354, Santiago, Metropolitana de Santiago
  - Local Institution - 350, Santiago, RM
  - Local Institution - 355, Recoleta, Santiago Metropolitan
  - Local Institution - 353, Santiago, Santiago Metropolitan
  - Local Institution - 352, Santiago, Santiago Metropolitan
- China (9):
  - Local Institution - 653, Beijing, Beijing Municipality
  - Local Institution - 657, Guangzhou, Guangdong
  - Local Institution - 655, Zhengzhou, Henan
  - Local Institution - 660, Wuhan, Hubei
  - Local Institution - 662, Shenyang, Liaoning
  - Local Institution - 663, Shenyang, Liaoning
  - Local Institution - 650, Shanghai, Shanghai Municipality
  - Local Institution - 651, Tianjin, Tianjin Municipality
  - Local Institution - 659, Guangzhou
- Denmark (3):
  - Local Institution - 602, Aarhus
  - Local Institution - 601, Copenhagen
  - Local Institution - 603, Vejle
- France (9):
  - Local Institution - 407, Bordeaux
  - Local Institution - 403, Créteil
  - Local Institution - 406, Lille
  - Local Institution - 409, Montpellier
  - Local Institution - 405, Paris
  - Local Institution - 402, Pierre-Bénite
  - Local Institution - 404, Rouen
  - Local Institution - 408, Toulouse
  - Local Institution - 401, Villejuif
- Israel (3):
  - Local Institution - 150, Jerusalem
  - Local Institution - 151, Petah Tikva
  - Local Institution - 152, Ramat Gan
- Italy (5):
  - Local Institution - 501, Bergamo
  - Local Institution - 504, Bologna
  - Local Institution - 503, Milan
  - Local Institution - 502, Napoli
  - Local Institution - 506, Pavia
- South Korea (4):
  - Local Institution - 553, Busan
  - Local Institution - 551, Seoul
  - Local Institution - 550, Seoul
  - Local Institution - 552, Seoul
- Spain (6):
  - Local Institution - 306, Badalona (Barcelona)
  - Local Institution - 301, Barcelona
  - Local Institution - 302, Madrid
  - Local Institution - 304, Madrid
  - Local Institution - 303, Málaga
  - Local Institution - 305, Salamanca
- United Kingdom (2):
  - Local Institution - 802, Edinburgh Scotland
  - Local Institution - 803, Southhampton

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT03930953.html